CLINICAL TRIAL: NCT05665803
Title: Comparative Evaluation of Instrumentation Time, Obturation Quality, and Child's Behavior Using Pediatric Rotary Versus Hand (Flare) File Systems in Treatment of Primary Molars: a Split Mouth Randomized Clinical Trial
Brief Title: Comparative Evaluation of Instrumentation Time Using Pediatric Rotary Versus Hand (Flare) File Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Wafik Ismael Mohamed, Assistant lecturer, department of pediatric dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pediatric rotary files
Record Dates: First submitted 2022-12-06; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Instrumentation Time
Keywords: Rotary files; Manual flare files

STUDY DESIGN:
Intervention Model Description: Split mouth RCT
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric rotary files (Experimental): Biomechanical preparation will be done using pediatric rotary file system (Kedo-SG blue file system). D1 and E1 files will be used at 300 rpm and 2.4 N/cm torque.
  Interventions: Procedure: Pediatric rotary files
- Manual flare files (Active Comparator): Biomechanical preparation will be done using manual flare files (Mani) No. 15-35.
  Interventions: Procedure: Manual flare files

INTERVENTIONS:
Procedure: Pediatric rotary files — Mechanical preparation of primary tooth canals with pediatric rotary files
  Arms: Pediatric rotary files
Procedure: Manual flare files — Mechanical preparation of primary tooth canals with manual flare files
  Arms: Manual flare files

SUMMARY:
The study will be conducted to evaluate instrumentation time, obturation quality, and child's behavior using pediatric rotary versus hand flare file systems in treatment of primary molars.

DETAILED DESCRIPTION:
Statement of the problem:

Pulpally affected primary teeth is a common problem in children due to lower mineralization, the presence of large pulp chamber with high pulp horns, and thin layers of enamel and dentin .

Manual files system is usually used for management of pulpally affected primary molars. This system has shown through the past years an acceptable clinical success rate but it also have many problems such as long visit time affecting the child behavior and causing fatigue to the dentist, difficulty in dealing with thin and curved canals due to limited flexibility of manual files causing incomplete removal of pulp tissue, and also difficulty in the determination of the actual working length due to the presence of physiologic and pathologic root resorption.

Rationale for conducting the research:

Pulp therapy in primary molars becomes compromised sometimes after delayed treatment due to dental neglect of children till caries progression to the pulp leading to severe symptoms associated with excessive pulp inflammation, root resorption, or periradicular bone resorption with a less favorable prognosis for conventional endodontic therapy. In the current era, a new perspective which is less time consuming with an acceptable success rate could be a spark of hope for the pediatric patient as well as the dentists.

Many studies were done comparing manual vs pediatric rotary files but without definitive conclusion. So further studies should be done with higher sample size to determine the superiority of one system over the other.

Benefits for the practitioner:

* Providing new and alternative treatment options.
* Shorter instrumentation time.
* Less fatigue.
* Better preparation of the canal.

Benefits for the patient:

* A faster and easier process leading to a more efficient dental procedure which could develop better outcomes in terms of success.
* Improvement in patient as well as parent satisfaction.

Benefits for community:

* Using alternative technique that can be faster, with a better success rate.
* To boost overall oral health.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Cooperative children.
* 4-6 years old children.
* Children who will attend follow up.

Teeth:

* Bilateral lower second primary molars.
* Pulpally involved molars indicated for pulpectomy.

Exclusion Criteria:

Children:

* Children with physical or emotional alteration.
* Children with systemic diseases.
* Children of parents who don't accept to participate in the study.

Teeth:

* Teeth with more than 1/3 of root resorption.
* Teeth with pathological mobility.
* Necrotic teeth with periapical or furcal lesions.
* Non restorable teeth.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 23 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Instrumentation time | during procedure
  Continuous outcome measured by digital stopwatch in minutes

SECONDARY OUTCOMES:
Child's behaviour | during procedure
  Using modified frankel scale from 1-5, where scale 1 has the worse behavior and scale 5 has the best behavior
Postoperative pain | 7 days
  Binary outcome reported by telephone call to the parents
Tenderness to percussion | 1 year
  Binary outcome measured by percussion test using back of the dental mirror
Pain on biting | 1 year
  Binary outcome reported by the patient at biting
Swelling/ fistula / sinus tract | 1 year
  Binary outcome measured with visual examination of the patient
Mobility | 1 year
  Binary outcome measured by mobility test using back of the two dental mirrors
Internal or external root resorption | 1 year
  Binary outcome using digital radiograph
Furcation involvement or periapical radiolucency | 1 year
  Binary outcome using digital radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Manal A Elsayed, Professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No
Data may be provided upon request